CLINICAL TRIAL: NCT01301001
Title: A Controlled Trial of Gabapentin in Vulvodynia: Biological Correlates of Response
Brief Title: A Trial of Gabapentin in Vulvodynia: Biological Correlates of Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 10-00985-FB CSBrown Vulvodynia
Record Dates: First submitted 2010-05-13; First posted 2011-02-23 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2016-04

CONDITIONS: Vulvodynia
Keywords: Vulvodynia
MeSH Terms: conditions — Vulvodynia | interventions — Sugars; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo oral capsule (Placebo Comparator): Placebo capsule daily in first intervention period and Gabapentin capsule 3000 mg daily in in second intervention (after washout period)
  Interventions: Drug: Placebo oral capsule; Drug: Gabapentin
- Gabapentin (Active Comparator): Gabapentin capsule 3000 mg daily in first intervention period and Placebo capsule in second intervention (after washout period)
  Interventions: Drug: Placebo oral capsule; Drug: Gabapentin

INTERVENTIONS:
Drug: Placebo oral capsule — Placebo 2 capsules am and 3 capsules pm
  Other Names: Sugar pill
Drug: Gabapentin — Gabapentin 1200 mg am and 1800 mg pm
  Other Names: Gralise 600 mg capsule

SUMMARY:
The Specific aims of this project are to (1) test the prediction that pain from tampon insertion (primary outcome measure) is lower in PVD patients when treated with gabapentin compared to when treated with placebo. Secondary outcome measures include intercourse pain and 24-hour pain and (2)perform a mechanism-based analysis of gabapentin effectiveness, and to gain insight into the underlying pathophysiology of subtypes of PVD that may lead to more specific treatment options.

DETAILED DESCRIPTION:
This is a 18-week, randomized, double-blind, placebo-controlled, two-treatment, two-period crossover design, where 120 women between 18 of age and older who report insertional dyspareunia, pain with tampon insertion, and tenderness localized to the vulvar vestibule will be enrolled in the study. Electronically entered daily diaries will be used to determine if pain is lower in PVD subjects when treated with gabapentin (up to 3600 mg/d) compared to when treated with placebo. Biological measurements will include assessment of allodynia and hyperalgesia from capsaicin administration, muscle tension using a vaginal pressure algometer, number of tender points by clinical examination, and changes in blood pressure, pulse and heart rate variability. . The Long-range goals of this project are to explicate the underlying pathophysiologic mechanisms of PVD, and to use this knowledge to create evidence-based differential diagnoses of subtypes of PVD and to individualize treatments for each subtype. The immediate goal is to conduct a multicenter, randomized controlled trial (RCT) of gabapentin treatment for PVD, and which will also provide critical data on a new PVD-testing and response paradigm, as well as on characteristics that may define subtypes of PVD. Gabapentin, an anticonvulsant with analgesic, anxiolytic, and antispasmotic effects, was selected because of its efficacy in treating other neuropathic pain conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are 18 years of age and older, as long as no vaginal atrophy is present. If vaginal atrophy is present, then topical hormone replacement can be provided for a minimum of 6 weeks and then she must be re-screened to be eligible,
2. Greater than 3 continuous months of insertional (entryway) dyspareunia, pain to touch, or both with tampon insertion (modified 'Friedrich's Criteria', and
3. an average pain level of "4" or greater on the 11-point tampon test (0 = no pain at all; 10 = worse pain ever) during the 2-week screening period must be exhibited.

(One tampon will be inserted each week). 4.) Must report pain with the "Tampon Insertion Pain" Test at visit 1

Exclusion Criteria:

1. Other vulvar conditions, including dermatoses, vulvitis, vulvar papillomatosis, or atrophic vaginitis (presence of a maturation index)
2. previous vestibulotomy
3. active vaginal infection (positive Affirm ™ VPIII microbial identification test)
4. pregnancy or at risk for pregnancy and not using a reliable birth control method for at least 3 months prior to entering the study
5. any unstable medical condition, including renal impairment (creatinine clearance of ≤60 mL/min, BUN > 30mg/dL, serum creatinine > 2 mg/dL), significant hematological disease (leukopenia [WBC < 3.0 x 10-3µl, leukocytosis [WBC >20.0 x 10-3μl], neutropenia [ABS < 1.50 x 10-3 μl, <20%]), (thrombocytopenia [platelets < 100,000 μl], anemia [HCT < 27%, HBG <8 g/dL, RBC <3 x 10-6]), cardiovascular disease (cardiac conduction disturbance, CHF, hypertension [140/90]), hepatic insufficiency (serum AST, ALT, or ALP ≥ 3 times upper limit of normal), neurological disorder (seizures, syncopal episodes, peripheral neuropathy, severe pain other than that caused by vulvodynia), autoimmune disease, or respiratory illness
6. psychiatric disorder, including history of major depressive disorder or substance abuse disorder within the past 6 months, a score of > 12 on the depression subscale of the Hospital Anxiety and Depression Scale (HADS), indicting a major depressive episode (35,36), a serious risk of suicide, or lifetime history of psychosis, hypomania or mania
7. multiple allergies
8. use of benzodiazepines, opiates, muscle relaxants, tricyclic antidepressants (TCAs), serotonin-norepinephrine reuptake inhibitors (SNRIs) or CNS stimulants (including methylphenidate, amphetamine dextroamphetamine) within 2 weeks of randomization and during the study
9. use of certain herbal agents within 2 weeks of randomization and during the study, including ginkgo biloba, evening primrose, St. John's Wort, Valerian, kava kava)
10. topical lidocaine use
11. Subjects, who are diagnosed with coexisting vaginismus, fibromyalgia and/or interstitial cystitis, must have greater vulvar pain than their coexisting conditions or they will not be eligible for study participation
12. Subject who have previously taken gabapentin or Lyrica but discontinued the medication due to side effects are not eligible
13. Subjects with active infections (Candida, BV, trichomonas, chlamydia, GC and HSV via Affirm/culture) must be treated and re-screened to eligible for participation
14. Subjects with 10% or greater parabasal cells and/or vaginal atrophy can be provided with topical hormone replacement for a minimum of 6 weeks and then must be re-screened to be eligible
15. Subjects who have had gastric bypass surgery are ineligible for study participation due to drug absorption problems
16. HPV/abnormal Pap is not exclusionary
17. Ongoing counseling and/or physical therapy is not exclusionary
18. Subjects who report signs of mixed Vulvodynia (spontaneous/provoked, localized, generalized) during prescreening will not be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace S Brown, MSN, PharmD, Principal Investigator — University of Tennessee; David C Foster, M.D., Principal Investigator — University of Rochester; Gloria A Bachmann, M.D., Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (3):
- United States (3):
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of Rochester School of Medicine and Dentistry, Rochester, New York
  - Clinical Research Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Brown CS, Bachmann GA, Wan J, Foster DC; Gabapentin (GABA) Study Group. Gabapentin for the Treatment of Vulvodynia: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jun;131(6):1000-1007. doi: 10.1097/AOG.0000000000002617. PMID 29742655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between August 8, 2012 and January 19, 2016 from three academic centers.
Pre-assignment Details: 230 women were screened, 89 met entry criteria and 66 completed the trial. Of the 141 patients who were excluded prior to randomization, 16 decided not to participate in the trial,101 did not meet inclusion criteria, and 24 did not return for randomization.
Groups:
- Placebo First, Then Gabepentin: Placebo capsule daily in first intervention period and Gabapentin capsule 3000 mg daily in in second intervention (after washout period)
  Placebo oral capsule: Placebo 2 capsules am and 3 capsules pm
  Gabapentin: Gabapentin 1200 mg am and 1800 mg pm
- Gabapentin First, Then Placebo: Gabapentin capsule 3000 mg daily in first intervention period and Placebo capsule in second intervention (after washout period)
  Placebo oral capsule: Placebo 2 capsules am and 3 capsules pm
  Gabapentin: Gabapentin 1200 mg am and 1800 mg pm
Period: First Intervention
Arm/Group | Placebo First, Then Gabepentin | Gabapentin First, Then Placebo
Started | 44 | 45
Completed | 34 | 36
Not Completed | 10 | 9
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Adverse Event | 5 | 0
Not completed — Protocol Violation | 0 | 1
Period: Washout (2 Weeks)
Arm/Group | Placebo First, Then Gabepentin | Gabapentin First, Then Placebo
Started | 34 | 36
Completed | 34 | 36
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo First, Then Gabepentin | Gabapentin First, Then Placebo
Started | 34 | 36
Completed | 30 | 36
Not Completed | 4 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: 44 subjects were randomized to Placebo First and 45 subjects were randomized to Gabapentin First
Arm/Group | All Study Participants
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.54 (2.30)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 89
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 58
  White | 30
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 89

OUTCOME MEASURES:

1. Primary Outcome: Tampon Test Pain Intensity
Description: Tampon pain on a 11-point Numeric Rating Scale (0 = no pain at all; 10 = worse pain ever). One tampon was inserted each week. Tampon pain was assessed during last week of maintenance phase (7 days).
Time Frame: Week 6 for each treatment arm
Population: Intention to Treat
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Placebo: 2 capsules am and 3 capsules pm
- Gabapentin: 2 capsules (1200 mg) am and 3 capsules (1800 mg) pm
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 89 | 89
units on a scale | 4.29 [3.37 to 5.22] | 3.96 [3.03 to 4.89]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin; Test type: Superiority; p = 0.07, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.7 to 0.0]

2. Secondary Outcome: Coital Pain
Description: Coital pain on an 11-point Numeric Rating Scale (0 = no pain at all; 10 = worse pain ever), assessed after each sexual intercourse event. The number of sexual intercourse events was averaged during final week of each treatment arm.
Time Frame: Week 6 of each treatment arm
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Gabapentin: 1200 mg am and 1800 mg pm
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 89 | 89
units on a scale | 3.97 [2.50 to 5.44] | 3.85 [2.36 to 5.34]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin; Test type: Superiority; p = 0.76, Mixed Models Analysis; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.9 to 0.6]

3. Secondary Outcome: Vulvodynia Pain
Description: Overall vulvodynia pain on an 11-point Numeric Rating Scale (0 = no pain at all; 10 = worse pain ever). Pain was assessed daily during the last week of treatment. Daily scores were averaged.
Time Frame: Week 6 for each treatment arm
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 89 | 89
units on a scale | 2.88 [1.99 to 3.76] | 2.71 [1.82 to 3.59]
Statistical Analysis 1: Comparison: Placebo vs Gabapentin; Test type: Superiority; p = 0.36, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.2]

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Definition of adverse events is the same as clinicaltrials.gov
Groups:
- Gabapentin: 2 capsules (1200 mg) am and 3 capsules (1800) mg pm
Arm/Group | Placebo | Gabapentin
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/89
Serious Adverse Events (participants affected / at risk) | 1/89 | 0/89
Other Adverse Events (participants affected / at risk) | 20/89 | 31/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=89) | Gabapentin (N=89)
unstable angina and malignant hypertension (Cardiac disorders) | 1 (1) | 0 (0)
asthma with acute exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cluster headache (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=89) | Gabapentin (N=89)
Dizziness (Nervous system disorders) | 3 (3) | 9 (17)
Fatigue (Nervous system disorders) | 1 (1) | 5 (7)
Headache (Nervous system disorders) | 5 (7) | 7 (15)
Somnolence (Nervous system disorders) | 4 (4) | 7 (7)
Rhinitis (Infections and infestations) | 4 (4) | 10 (14)
Nausea (Gastrointestinal disorders) | 3 (4) | 8 (13)
Bacterial Vaginosis (Infections and infestations) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes